CLINICAL TRIAL: NCT01792986
Title: Preparatory Study to Determine Which Risk Markers May be Reduced by Fasting and Should be Evaluated in a Future Randomized Trial
Brief Title: The Fasting II Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Intermountain Research and Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1024469
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2013-07

CONDITIONS: Diabetes; Metabolic Diseases
Keywords: Diabetes; Fasting; Pre-diabetes; Hemoglobin A1C
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Diseases; Fasting; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- water-only 24-hour fasting once per week for 6 weeks (Other)
  Interventions: Behavioral: water-only 24-hour fasting once per week for 6 weeks

INTERVENTIONS:
Behavioral: water-only 24-hour fasting once per week for 6 weeks

SUMMARY:
This study will determine whether an intensive fasting protocol alters hemoglobin A1c measurements or other markers of metabolic and cardiovascular risk by performing a 5-week clinical trial of fasting among 12 pre-diabetic individuals or diabetics whose disease is controlled by diet. Participants will undergo a 5-week intervention of once-per-week 24-hour water-only fasting, including at baseline and at the end of the week for each week of the study (a total of 6 24-hour fasts).

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female, ≥30 and <70 years of age.
2. Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures.
3. Prior evidence of pre-diabetic state, with one of the following:

   1. Pre-diabetic with a measured hemoglobin A1c (HbA1c) ≥6.0% or fasting glucose >100 mg/dL without a clinical diabetes diagnosis
   2. Clinically-diagnosed type II diabetic with HbA1c ≥6.0% or fasting glucose ≥110 mg/dL and whose disease is controlled by diet alone.
4. Evidence of metabolic syndrome by having at least 3 of the following 5 criteria:

   1. Fasting glucose level >100 mg/dL.
   2. Blood pressure ≥135 mmHg systolic or ≥85 mmHg diastolic, or use of an antihypertensive medication.
   3. High-density lipoprotein cholesterol <40 mg/dL in males or <50 mg/dL in females.
   4. Triglycerides ≥150 mg/dL or use of a cholesterol-lowering medication.
   5. Waist circumference >40 inches (102 cm) for males or >35 inches (88 cm) for females (or body mass index >25 kg/m2).

Exclusion Criteria:

1. Pregnant and/or lactating women and women of child bearing potential who are not using acceptable means of contraception. Women of childbearing potential must be using adequate measures of contraception (as determined by the Principal Investigator) to avoid pregnancy and should be highly unlikely to conceive during the study period. Women of childbearing potential must have a negative pregnancy test at screen.
2. Diabetics taking any of the following anti-diabetic medications: insulin, metformin, thiazolidinediones, sulfonylureas, alpha-glucosidase inhibitors, meglitinides, or incretins.
3. Prior experience with fasting more than once per month (for 20 hours or more), on average during the last year.
4. Very low body mass index (BMI) (<18.5 kg/m2) or high BMI (>40 kg/m2).
5. Individuals who are nutritionally compromised, as assessed by the Principal Investigator.
6. Any immunodeficiency or prior solid organ transplantation or renal disease.
7. Participation in any other clinical trials involving investigational or marketed products within 30 days prior to entry in the study.
8. Other conditions that in the opinion of the Principal Investigator may increase risk to the subject and/or compromise the quality of the clinical trial.

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Horne, PhD, MPH, Principal Investigator — Intermountain Health Care, Inc.
Locations (2):
- United States (2):
  - Intermountain Medical Center, Murray, Utah
  - Intermountain Medical Center, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Water-only 24-hour Fasting Once Per Week for 6 Weeks: water-only 24-hour fasting once per week for 6 weeks
Period: Overall Study
Arm/Group | Water-only 24-hour Fasting Once Per Week for 6 Weeks
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Water-only 24-hour Fasting Once Per Week for 6 Weeks
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Difference in Mean Glucose Level Between Baseline and the End of the Sixth Week.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Water-only 24-hour Fasting Once Per Week for 6 Weeks
Number analyzed (Participants) | 12
mg/dL
  Baseline | 104.7 (17.7)
  6-week | 104.5 (18.8)

2. Secondary Outcome: Difference in Weight Between Baseline and the End of the Sixth Week
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Water-only 24-hour Fasting Once Per Week for 6 Weeks
Number analyzed (Participants) | 12
kg
  Baseline | 92.5 (11.3)
  6-week | 90.9 (11.1)

3. Secondary Outcome: Difference in Low-density Lipoprotein Cholesterol (LDL-C) Between Baseline and the End of the Sixth Week.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Water-only 24-hour Fasting Once Per Week for 6 Weeks
Number analyzed (Participants) | 12
mg/dL
  Baseline | 100.9 (38.1)
  6-week | 87.8 (27.4)

4. Secondary Outcome: Difference in Human Growth Hormone (HGH) Between Baseline and the End of the Sixth Week.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Water-only 24-hour Fasting Once Per Week for 6 Weeks
Number analyzed (Participants) | 12
ng/mL
  Baseline | 0.69 (1.04)
  6-week | 0.51 (0.53)

5. Secondary Outcome: Difference in Red Blood Cell Count Between Baseline and the End of the Sixth Week.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: trillion cells/L
Arm/Group | Water-only 24-hour Fasting Once Per Week for 6 Weeks
Number analyzed (Participants) | 12
trillion cells/L
  Baseline | 4.82 (0.34)
  6-week | 4.78 (0.35)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Water-only 24-hour Fasting Once Per Week for 6 Weeks
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes